CLINICAL TRIAL: NCT00946556
Title: Examining the Ability of HSV2 Therapy to Reduce HIV Target Cell Numbers in the Cervix.
Brief Title: Examining the Ability of Herpes Simplex Virus Type 2 (HSV2) Therapy to Reduce HIV Target Cell Numbers in the Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Rupert Kaul, Dr., University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HET-85518
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Herpes Simplex Type Two Infection; HIV Infections
Keywords: herpes simplex virus type 2; HIV; genital immunology; CD4+ T cell; valacyclovir; HIV seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will be assigned 2 months of placebo or active drug, with an intervening one month washout period.
  Interventions: Drug: Valacyclovir; Drug: Placebo
- Valacyclovir (Experimental): Participants will be assigned 2 months of placebo or active drug, with an intervening one month washout period.
  Interventions: Drug: Valacyclovir; Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — 1g po od for 2 months
Drug: Placebo — Placebo po od for 2 months

SUMMARY:
Herpes simplex virus type 2 (HSV2), the most common cause of genital herpes, increases a woman's risk of HIV acquisition from 3-6 fold, perhaps because HSV2-infected women have increased numbers of HIV "target cells" (CD4 T cells and dendritic cells) in the cervical mucosa. However, recent clinical trials showed no impact of HSV2 suppression on HIV acquisition rates. The reasons for this negative result are unclear. The investigators propose to examine the effect of valacyclovir (a widely used herpes medication) treatment on cervical immunology and HIV target cells in the cervix. The study will take the form of a randomized, double-blind, placebo-controlled crossover trial. Primary endpoints will be (1) the number of CD4 T cells on a cervical cytobrush and (2) the number of immature dendritic cells per cervical cytobrush.

ELIGIBILITY:
Inclusion Criteria:

* Female
* HSV2 infected

Exclusion Criteria:

* HIV infected
* Pregnant
* Taking HSV2 therapy
* Current/recent (past 3 months) genital infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of CD4+ T cells on a cervical cytobrush. | Monthly intervals for 5 months

SECONDARY OUTCOMES:
Number of immature dendritic cells on a cervical cytobrush | Monthly intervals for 5 months
Proinflammatory cytokine/chemokine levels in cervicovaginal secretions | Monthly intervals for 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Kaul, MD/PhD, Principal Investigator — University of Toronto
Locations (1):
- Women's Health In Women's Hands, Toronto, Ontario, Canada

REFERENCES:
- [Background] Rebbapragada A, Wachihi C, Pettengell C, Sunderji S, Huibner S, Jaoko W, Ball B, Fowke K, Mazzulli T, Plummer FA, Kaul R. Negative mucosal synergy between Herpes simplex type 2 and HIV in the female genital tract. AIDS. 2007 Mar 12;21(5):589-98. doi: 10.1097/QAD.0b013e328012b896. PMID 17314521
- [Derived] Yi TJ, Shannon B, Chieza L, Su D, Saunders M, Tharao W, Huibner S, Remis R, Raboud J, Kaul R. Valacyclovir therapy does not reverse herpes-associated alterations in cervical immunology: a randomized, placebo-controlled crossover trial. J Infect Dis. 2014 Sep 1;210(5):708-12. doi: 10.1093/infdis/jiu163. Epub 2014 Mar 23. PMID 24664172